CLINICAL TRIAL: NCT03786250
Title: Comprehensive Geriatric Assessment in Emergency Department. Impact on Health and Patient Flows
Brief Title: Comprehensive Geriatric Assessment in an Emergency Department
Acronym: CGA_ED
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Fundació Mutuam Conviure (Unknown)
Responsible Party: Sponsor
Other Study IDs: IIBSP-AGI-2017-14
Record Dates: First submitted 2018-12-11; First posted 2018-12-26 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Emergencies; Aging; Geriatric Assessment; Patient Discharge
Keywords: Emergency department; Older; Frailty
MeSH Terms: conditions — Emergencies; Frailty | interventions — Geriatric Assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Geriatric Assessment — Systematic screening of delirium, prevention of delirium, early treatment, pain management with scales adapted to chronicity, conciliation of medication to emergency discharge, among others.
  Other Names: CGA

SUMMARY:
Purpose Frailty and multi-morbidity have been associated with increased pressure on Emergency Departments (ED), higher hospital admissions and more risks for patients arising from the ED stay. The advantages of developing specific attention to frailty in ED have been highlighted. The benefits of these approaches are related to patients but also to organizations. The aim is to present how a Program of Care for Frailty (PCF) in an ED impacts on patient health and flows.

Objective is to analyze the clinical impact of Comprehensive Geriatric Care (CGA) in the Emergency Department (ED) and on patient flows Setting: A tertiary, teaching, 550-bed urban hospital, with 80,000 adult patients/year ED attendances (43%≥65 years). Two periods are compared: First period (before CGA implantation) del 01/04/2016 - 15/04/2016 and second period (after) 01/04/2017 - 15/04/2017

DETAILED DESCRIPTION:
Purpose Frailty and multi-morbidity have been associated with increased pressure on Emergency Departments (ED), higher hospital admissions and more risks for patients arising from the ED stay. The advantages of developing specific attention to frailty in ED have been highlighted. The benefits of these approaches are related to patients but also to organizations. The aim is to observe how a Program of Care for Frailty (PCF) in an ED impacts on patient health and flows.

Objective

1. Analyze the clinical impact of Comprehensive Geriatric Care (CGA) in the Emergency Department (ED).
2. Analyze the impact on patient flows following the implementation of a Comprehensive Geriatric Assessment in the Emergency Department (ED).

Methods Setting: A tertiary, teaching, 550-bed urban hospital, with 80,000 adult patients/year ED attendances (43%≥65 years).

First period (before CGA implantation) del 01/04/2016 - 15/04/2016 and second period (after) 01/04/2017 - 15/04/2017 Intervention: In the second period, the AGI was carried out by the emergency medical teams. It basically consists of care adapted to the special needs of geriatric patients, with systematic screening of delirium, delirium prevention, early treatment, pain management with scales adapted to chronicity, conciliation of medication to discharge from the emergency department, among others A comparison will be made of health outcomes and patient flows in ED: direct discharge, admission to emergency observation unit, admission to short stay unit, transfer to intermediate hospital, admission, admission to critical care area, death, time spent in the Emergency Department (ED) and in intermediate hospital, mortality during admission at one and six months, re-entry or reconsultation in the Emergency Department at 30 days and six months will be measured.

ELIGIBILITY:
Inclusion Criteria:

* All patients older than 65 years attended in the ED

Exclusion Criteria:

* None

Ages: 18 Years to 115 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients older than 65 years, attended in ED during the study periode.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with delirium | From date of admission until discharge, assessed up to 30 days

SECONDARY OUTCOMES:
Number of patients with pain correctly treated | From date of admission until discharge, assessed up to 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided